CLINICAL TRIAL: NCT03202771
Title: Home Versus Office Biofeedback Training for Dyssynergic Defecation
Brief Title: Randomized Controlled Trial of Home Versus Office Biofeedback for Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2RO1-DK057-100-06A
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-06

CONDITIONS: Constipation; Dyssynergia
MeSH Terms: conditions — Constipation; Ataxia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Biofeedback Therapy (Experimental): Patients will use home biofeedback device to practice their maneuvers taught by the nurse.
  Interventions: Device: Home Biofeedback Therapy
- Office Biofeedback Therapy (Active Comparator): Patients will get regular office biofeedback therapy with an anal probe inserted while a nurse runs through the exercise session together.
  Interventions: Other: Office Biofeedback Therapy

INTERVENTIONS:
Device: Home Biofeedback Therapy — Patients will be taught how to use the home-trainer in a single lab session. Then we will place a reusable, dual sensor, probe into their rectum. The probe is connected to a hand- held pressure monitor displaying the patient's response. Next, the clothed patient will be asked to sit on a commode, and attempt 15 bearing down maneuvers. When the anal sphincter pressure decreases more lights go on. If the patient cannot relax then fewer lights go on. Thus, the number of lighted lights gives instant feedback about their performance. Patients will get a 20-minute tape recording for home use. Patients will be asked to insert the probe at least twice daily and each time practice at least 15 bearing down maneuvers; a daily log will be kept. At 4 and 8 weeks, they will return for follow up. Based on their progress, new targets will be set by adjusting the device's sensitivity.
  Arms: Home Biofeedback Therapy
Other: Office Biofeedback Therapy — A monitor screen will provide visual feedback by showing changes in pressure activity. First patients will be taught abdominal muscle coordination exercise to improve the pushing effort during defecation. Here, patients are taught how to distend the abdomen by inhaling slowly and then holding their breath for at least 15 seconds and to practice this for 20 minutes, twice a day. Thereafter, patients will be asked to attend the motility laboratory, biweekly for up to 6 training sessions. Biofeedback Therapy (BT) will be performed by a 3-sensor manometry probe. The clothed patient will be seated on a commode in front of a monitor. The physician/nurse therapist will give verbal feedback by either complimenting the patient for performing a correct maneuver or rectifying any errors. Each 60 minute treatment session will comprise of the following maneuvers:
  Arms: Office Biofeedback Therapy

SUMMARY:
Test the Efficacy of Home Biofeedback Training: Currently, biofeedback requires a skilled therapist and sophisticated equipment and is not widely available. The investigators designed and tested a novel home biofeedback device and predict that home training will be as effective as office biofeedback therapy. Our specific aims are to perform a randomized controlled trial of 100 subjects with dyssynergic defecation to investigate:

(A) Whether a self-administered, home-biofeedback training program with a new portable device is as effective as office-based biofeedback therapy in improving i) physiology- dyssynergia (defecation index), and ability to expel simulated stool, and ii) symptomatology- satisfaction with bowel function, number of complete spontaneous bowel movements, stool consistency, straining and quality of life.

(B) Whether home-training is more cost-effective than office-based biofeedback training.

DETAILED DESCRIPTION:
Study Protocol: Patients will be randomized to receive either office-based biofeedback therapy or home-based biofeedback training, in addition to the standard treatment described below.

Randomization procedures: The permuted blocks method will randomize patients for all study aims; this ensures approximate balance among the two treatment arms, while making it unlikely that investigators will predict the next treatment assignment. The study statistician will prepare sequentially numbered sealed envelopes containing the treatment assignment. Thus the next treatment assignment cannot be read without opening the envelope. If a patient is deemed eligible, and agrees to participate, after signing the informed consent, the investigator will open the next envelope to determine the treatment assigned to that patient.

Standard Treatment: The patient will be seen by one of the gastroenterologists and receive instructions regarding their problem and advice on exercises, timed toilet training, laxatives, diet and fluid intake. Written materials will be given to each patient and the study coordinator will reinforce the information.

Timed-toilet training: This consists of educating the patient regarding the anatomy and physiology of the pelvic floor and diaphragmatic breathing technique. They will be advised to attempt a bowel movement twice a day, 30 minutes after meals and strain for five minutes and push at a level of 5-7/10.

Laxatives: Patients will be asked to use 500 mg magnesium gluconate, 2-3 tablets/day or Milk of Magnesia 1-3 tablespoons daily. If intolerant, they will be advised to use bisacodyl (1-2 daily) or sennokot (1-2 daily), but to titrate the dose. Patients will be asked to refrain from using digital maneuvers and enemas. Rescue medications will include bisacodyl suppositories (no BM for 48 hrs) or enema (no BM for 72 hours). If bowel movement is regular i.e. soft stool >3/week, they will be asked to reduce the laxative dose by 1/3rd.

Diet: Based on a three-day prospective food diary, patients will get advice by the GCRC dietician. The recommendations will include the advice to eat 5 servings of fruits and vegetables per day, and 25 g dietary fiber from natural foods, and consume ~30% of calories from fat. Three-day food records, obtained at baseline, and at 4, 8 and 12 weeks, will assess dietary compliance. Subjects will get a diet report to reinforce adherence.

Office Biofeedback (Neuromuscular conditioning) Treatment- The aim of biofeedback will be to establish a normal pattern of defecation and improve rectal sensation using visual/verbal biofeedback technique. A monitor screen will provide visual feedback by showing changes in pressure activity. First patients will be taught abdominal muscle coordination exercise to improve the pushing effort during defecation. Here, patients are taught how to distend the abdomen by inhaling slowly and then holding their breath for at least 15 seconds and to practice this for 20 minutes, twice a day. Thereafter, patients will be asked to attend the motility laboratory, biweekly for up to 6 training sessions. BT will be performed by a 3-sensor manometry probe. The clothed patient will be seated on a commode in front of a monitor. The physician/nurse therapist will give verbal feedback by either complimenting the patient for performing a correct maneuver or rectifying any errors. Each 60 minute treatment session will comprise of the following maneuvers:

Recto-Anal Coordination This maneuver's goal is to produce a coordinated movement that simultaneously increases the intra abdominal (intra rectal) pressure and relaxes the anal sphincter. First, the patient is educated about their abnormal tracing: A normal pattern is shown and they are encouraged to reproduce this. The patients' posture and breathing are continuously monitored and corrected and verbal reinforcement provided. If a patient consistently demonstrates normal rectoanal coordination, then they are asked to reproduce this without feedback. Approximately 15 bearing down maneuvers are performed at 1 minute intervals, some with and some without rectal balloon distention.

Simulated defecation: This is performed by placing a fecom (artificial stool) into the rectum. The patient is asked to sit on a commode and expel the fecom. Their movements, posture, and breathing techniques are corrected and feedback is provided. The therapist may assist the patient's effort by applying gentle traction to the fecom, while reinforcing their straining technique. The maneuver is repeated twice.

Assessment of Improvement: The number of training sessions will be customized for each patient (maximum 6). Training will be discontinued if a patient demonstrates during two consecutive training sessions, without feedback a) normal pattern of defecation in at least 50% of attempts, and b) at least 20% improvement in bowel satisfaction (VAS) (64). If these goals are not achieved, patients will be considered treatment failures.

Home Biofeedback Treatment: After getting advice on standard treatment and breathing exercises, patients will be taught how to use the home-trainer in a single lab session. Then the investigators will place a reusable, dual sensor, probe into their rectum. The probe is connected to a hand- held pressure monitor displaying the patient's response (Anatoner, Protech, Hyderabad, India). Next, the clothed patient will be asked to sit on a commode, and attempt 15 bearing down maneuvers. When the anal sphincter pressure decreases more lights go on. If the patient cannot relax then fewer lights go on. Thus, the number of lighted lights gives instant feedback about their performance. Patients will get a 20-minute tape recording for home use. Patients will be asked to insert the probe at least twice daily and each time practice at least 15 bearing down maneuvers; a daily log will be kept. At 4 and 8 weeks, they will return for follow up. Based on their progress, new targets will be set by adjusting the device's sensitivity. After 3-months, they will have a colonic transit, anorectal manometry and fecom expulsion study. Progress will be monitored through bi-weekly phone calls.

ELIGIBILITY:
Inclusion Criteria:

* During the previous year, all patients must have experienced or reported at least two of the following symptoms for at least three months and with 25% of bowel movements (when not taking laxatives):
* stool frequency of less than three/week,
* passage of hard stools,
* excessive straining,
* a feeling of incomplete evacuation,
* sensation of anorectal obstruction or blockage and
* use of manual maneuvers to facilitate defecations (e.g., digital evacuation).
* No evidence of structural disease (excluded by colonoscopy/ b. enema and metabolic problem by lab tests.
* Patients on stable doses of antidepressants without anticholinergic effects will be included.

Exclusion Criteria:

* Patients taking drugs that are constipating, (e.g.; calcium channel antagonists will either be excluded or drug discontinued)
* Patients with co-morbid illnesses; severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy.
* Neurologic diseases e.g.; head injury, epilepsy, multiple sclerosis, strokes, spinal cord injuries.
* Impaired cognizance (mini mental score of < 15) and/or legally blind.
* Pregnant or likely to conceive during the course of the study. Women with potential for pregnancy must be willing to use contraceptive measures during the study. Urinary pregnancy tests will be performed on such women prior to any radiologic procedures.
* Hirschsprung's disease.
* Alternating constipation and diarrhea.
* Ulcerative/Crohns colitis.
* Previous pelvic surgery, rectocele/bladder repair, radical hysterectomy, anal surgery.
* Rectal prolapse or anal fissure.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Presence of Dyssynergia | 3 months
  Dyssynergia pattern
Balloon Expulsion Time | 3 months
  Time it takes for a subject to expel a balloon that has been inserted into the rectum.
Number of Complete Spontaneous Bowel Movements | 3 months
  Number of how many bowel movements occur without using an aid to have a bowel movement.
Global Bowel Satisfaction | 3 months
  visual analog scale of symptoms

SECONDARY OUTCOMES:
Colon Transit | 3 months
  colon transit time

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao SSC, Go JT, Valestin J, Schneider J. Home Biofeedback for the Treatment of Dyssynergic Defecation: Does It Improve Quality of Life and Is It Cost-Effective? Am J Gastroenterol. 2019 Jun;114(6):938-944. doi: 10.14309/ajg.0000000000000278. PMID 31170114
- [Derived] Rao SSC, Valestin JA, Xiang X, Hamdy S, Bradley CS, Zimmerman MB. Home-based versus office-based biofeedback therapy for constipation with dyssynergic defecation: a randomised controlled trial. Lancet Gastroenterol Hepatol. 2018 Nov;3(11):768-777. doi: 10.1016/S2468-1253(18)30266-8. Epub 2018 Sep 18. PMID 30236904